CLINICAL TRIAL: NCT02596217
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising s.c. (Stage 1) and i.v. (Stage 2) Doses of BI 655066/ABBV-066 (Risankizumab) in Healthy Asian and Caucasian Male Volunteers (Double-blind, Randomized, Placebo-controlled Within Dose Groups)
Brief Title: Safety, Tolerability and Pharmacokinetics of BI 655066/ABBV-066 (Risankizumab) in Healthy Asian and Caucasian Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-513; 1311.16 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2015-08-12; First posted 2015-11-04 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: ABBV-066; BI 655066; risankizumab
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Stage 1 (low dose SC) (Experimental): Low dose administered by subcutaneous (SC) injection
  Interventions: Drug: ABBV-066
- Stage 1 (medium dose SC) (Experimental): Medium dose administered by subcutaneous (SC) injection
  Interventions: Drug: ABBV-066
- Stage 1 (high dose SC) (Experimental): High dose administered by subcutaneous (SC) injection
  Interventions: Drug: ABBV-066
- Stage 2 (low dose IV) (Experimental): Low dose administered by intraveneous (IV) infusion
  Interventions: Drug: ABBV-066
- Stage 2 (medium dose IV) (Experimental): Medium dose administered by intraveneous (IV) infusion
  Interventions: Drug: ABBV-066
- Stage 2 (high dose IV) (Experimental): High dose administered by intraveneous (IV) infusion
  Interventions: Drug: ABBV-066
- Placebo SC (Stage1) (Placebo Comparator): Placebo administered by subcutaneous (SC) injection
  Interventions: Drug: Placebo
- Placebo IV (Stage2) (Placebo Comparator): Placebo administered by intraveneous (IV) infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABBV-066 — SC injection
  Other Names: BI 655066; risankizumab
  Arms: Stage 1 (high dose SC); Stage 1 (low dose SC); Stage 1 (medium dose SC)
Drug: ABBV-066 — IV infusion
  Other Names: BI 655066; risankizumab
  Arms: Stage 2 (high dose IV); Stage 2 (low dose IV); Stage 2 (medium dose IV)
Drug: Placebo — SC injection (stage 1)
  Arms: Placebo SC (Stage1)
Drug: Placebo — IV infusion (stage 2)
  Arms: Placebo IV (Stage2)

SUMMARY:
Safety, tolerability and pharmacokinetics of single dose of BI 655066/ABBV-066 (risankizumab) in healthy Chinese, Japanese and Caucasian male volunteers.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects according to the investigator¿s assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
2. Chinese ethnicity, Japanese ethnicity, or Caucasian according to the following criteria:

   * Chinese; born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in china
   * Japanese; born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan
   * Caucasian
3. Age of 20 to 45 years (incl.)
4. BMI of 18.5 to 25 kg/m2 (incl.) for Chinese and Japanese subjects, BMI of 18.5 to 29.9 kg/m2 (incl.) for Caucasian subjects.
5. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.
6. Male subjects who agree to minimize the risk of female partners becoming pregnant by fulfilling any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:

   * Use of adequate contraception, e.g. any of the following methods plus condom: implants, combined oral or vaginal contraceptives, intrauterine device
   * Sexually abstinent
   * Vasectomised (vasectomy at least 1 year prior to enrolment)
   * Surgically sterilised (including hysterectomy)

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
2. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
3. Any evidence of a concomitant disease judged as clinically relevant by the investigator
4. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
5. Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
6. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
7. History of relevant orthostatic hypotension, fainting spells, or blackouts
8. Chronic or relevant acute infections including HIV, viral hepatitis and (or) tuberculosis or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold (or T-SPOT) test. Subjects with a positive QuantiFERON TB-Gold (or T-SPOT) test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment must have been initiated and maintained according to local country guidelines.
9. History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
10. Intake of biologic agents other than current study medication or drugs considered likely to interfere with the safe conduct of the study
11. Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
12. Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
13. Participation in another trial with an investigational drug within 90 days or 5 half-lives (whichever is greater) prior to planned administration of trial medication
14. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
15. Inability to refrain from smoking on specified trial days
16. Alcohol abuse (consumption of more than 30 g per day)
17. Drug abuse or positive drug screening
18. Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
19. Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
20. Inability to comply with dietary regimen of trial site
21. A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
22. A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
23. Have received any live bacterial or live viral vaccination in the 12 weeks prior to the date of screening. Subjects must agree not to receive a live bacterial or live viral vaccination during the study and up to 12 months after the last administration of study drug
24. Have received Bacille Calmette-Guerin (BCG) vaccination in the 12 months prior to the date of screening. Subjects must agree not to receive BCG vaccination during the study and up to 12 months after the last administration of study drug
25. Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with drug-related adverse events | Up to 144 days after screening

SECONDARY OUTCOMES:
Time from dosing to the maximum plasma concentration of the analyte in plasma (tmax) | Up to 144 days after randomization
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to time of the last quantifiable plasma concentration (AUC0-tz) | Up to 144 days after randomization
Maximum measured plasma concentration of the analyte in plasma (Cmax) | Up to 144 days after randomization
Terminal half-life of the analyte in plasma (t1/2) | Up to 144 days after randomization
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity) | Up to 144 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Boehringer Ingelheim Investigational Site, Tokyo, Sumida-ku, Japan
- Boehringer Ingelheim Investigational Site, Busan, South Korea

REFERENCES:
- [Derived] Thakre N, D'Cunha R, Goebel A, Liu W, Pang Y, Suleiman AA. Population Pharmacokinetics and Exposure-Response Analyses for Risankizumab in Patients with Active Psoriatic Arthritis. Rheumatol Ther. 2022 Dec;9(6):1587-1603. doi: 10.1007/s40744-022-00495-0. Epub 2022 Sep 30. PMID 36178584
- [Derived] Suleiman AA, Minocha M, Khatri A, Pang Y, Othman AA. Population Pharmacokinetics of Risankizumab in Healthy Volunteers and Subjects with Moderate to Severe Plaque Psoriasis: Integrated Analyses of Phase I-III Clinical Trials. Clin Pharmacokinet. 2019 Oct;58(10):1309-1321. doi: 10.1007/s40262-019-00759-z. PMID 31054118